CLINICAL TRIAL: NCT05523609
Title: Effect of Vitamin D and Calcium Supplementation on Letrozole-induced Musculoskeletal Side Effects in Breast Cancer Egyptian Patients
Brief Title: Vitamin D and Calcium Supplementation in Breast Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mai Abo Elyazeed Hassan Hamouda, Clinical Pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vitamin D and breast cancer
Record Dates: First submitted 2022-08-25; First posted 2022-08-31 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Cholecalciferol; Calcium

STUDY DESIGN:
Intervention Model Description: Forty breast cancer patients were included. They were divided into 2 equal groups: Control group received Letrozole only, and VitD/Ca group received Letrozole in addition to 2000 IU vitamin D3 and 1000 mg of calcium per day for 12 weeks. Baseline serum 25-hydroxy vitamin D concentrations were assayed and standard health assessment questionnaire was completed to assess the disability caused by musculoskeletal symptoms.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): 20 patients will receive Letrozole only for 12 weeks.
  Interventions: Drug: Letrozole 2.5mg
- VitD/Ca group (Experimental): 20 patients will receive Letrozole in addition to 2000 IU vitamin D3 and 1000 mg of calcium per day for 12 weeks.
  Interventions: Drug: Letrozole + vitamin D3 and calcium

INTERVENTIONS:
Drug: Letrozole 2.5mg — 20 patients will receive Letrozole only for 12 weeks
  Arms: Control Group
Drug: Letrozole + vitamin D3 and calcium — 20 patients will receive Letrozole in addition to 2000 IU vitamin D3 per day for 12 weeks.
  Arms: VitD/Ca group

SUMMARY:
This study aims at assessing the vitamin Dstatus in breast cancer patients who receive letrozole for more than two months and to evaluate effects of vitamin D3 and calcium supplementation on arthalgia caused by letrozole on these patients.

DETAILED DESCRIPTION:
Background: Vitamin D deficiency (< 10 ng/mL) and insufficiency (10-30 ng/mL) may contribute to musculoskeletal symptoms observed in patients taking letrozole. This study was undertaken to assess the vitamin D status in breast cancer patients who received letrozole for > 6 months and to evaluate the effects of vitamin D3 and calcium supplementation on them.

Methods: Forty breast cancer patients were included. They were divided into 2 equal groups: Control group received Letrozole only, and VitD/Ca group received Letrozole in addition to 2000 IU vitamin D3 and 1000 mg of calcium per day for 12 weeks. Baseline serum 25-hydroxy vitamin D concentrations were assayed and standard health assessment questionnaire was completed to assess the disability caused by musculoskeletal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed breast cancer patients.
* Postmenopausal hormone receptor positive.
* Patients receiving letrozole for more than two months
* Gender: Female.
* Age: ≥ 50 years old.

Exclusion Criteria:

* Patients with bone metastasis.
* History of renal stones.
* Serum calcium >11mg/L.
* Patients with renal insufficiency.
* Patients taking steroid hormone replacement therapy.
* Second Malignancy.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Osteocalcin level | 12 weeks
  Osteocalcin level at base line and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sahar K Hegazy, Professor, Study Director — Head of clinical Pharmacy Department
Locations (1):
- Tanta Cancer Center, Tanta, El-Gharbia, Egypt